CLINICAL TRIAL: NCT05755477
Title: Survey About the Relationship Beetween Allergic Rhinitis and Seasonal EOE Exacerbations: the Role of Respiratory Allergy in the EOE Etiopathogenesis
Brief Title: Survey About the Relationship Beetween Allergic Rhinitis and Seasonal EOE Exacerbations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nucera Eleonora (Other)
Responsible Party: Sponsor-Investigator, Nucera Eleonora, Professor, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Organization: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Other Study IDs: 3638
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Eosinophilic Esophagitis; Respiratory Allergy
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophilic esophagitis (EoE) is a chronic inflammatory esophagus disease that is presented in patients with a history of recurrent dysphagia.

EoE is closely related to other pathologies with an immuno-allergic etiopathogenesis such as atopic dermatitis (AD), IgE-mediated food allergy, allergic rhinitis and bronchial asthma.

While the importance of the correlation between diet and food allergy has been largely demonstrated, less is known about the exact role of sensitization to aerollergens in the progression and recrudescence of symptoms.

In support of this correlation there is evidence of a seasonal trend in the new diagnoses of EoE, of the possibility of the de-novo onset of the pathology following massive exposure to a specific aeroallergen and the demonstration that the degree of esophageal eosinophilia varies according to the climatic zone and the season of the year.

The detailed knowledge of this correlation could clarify some aspects of the etiopathogenesis and natural history of EoE, improve and personalize the clinical-diagnostic management of affected patients and provide new therapeutic targets.

Our aim is evaluating the possible existence of a correlation between the recrudescence of dysphagia symptoms and a specific month of the year and/or specific season.

DETAILED DESCRIPTION:
Eosinophilic esophagitis (EoE) is a chronic inflammatory esophagus disease that is presented in patients with a history of recurrent dysphagia.

EoE is closely related to other pathologies with an immuno-allergic etiopathogenesis such as atopic dermatitis (AD), IgE-mediated food allergy, allergic rhinitis and bronchial asthma.

While the importance of the correlation between diet and food allergy has been largely demonstrated, less is known about the exact role of sensitization to aerollergens in the progression and recrudescence of symptoms.

In support of this correlation there is evidence of a seasonal trend in the new diagnoses of EoE, of the possibility of the de-novo onset of the pathology following massive exposure to a specific aeroallergen and the demonstration that the degree of esophageal eosinophilia varies according to the climatic zone and the season of the year.

The detailed knowledge of this correlation could clarify some aspects of the etiopathogenesis and natural history of EoE, improve and personalize the clinical-diagnostic management of affected patients and provide new therapeutic targets.

It is a cross-sectional observational study and the aim is:

* evaluating the possible existence of a correlation between the recrudescence of dysphagia symptoms and a specific month of the year and/or specific season
* evaluating whether there is a statistically significant correlation between the anamnestic onset of the disease and the individual patient's sensitization to aeroallergens and the prevalence of respiratory allergy (rhinitis and allergic asthma) in patients with EoE.

All the patient should answer a questionnaire about the state of health over the year and according to the various pollen seasons

The questionnaire is made up of 18 questions which aim to investigate:

* anamnestic data (age, weight, height, clinical onset of the pathology);
* dysphagia symptomatology through modified DSQ (Dysphagia Symptom Questionnaire);
* rhinitis symptomatology SFAR (Score For Allergic Rhinitis);
* trend of exacerbations of dysphagia symptoms in the different months of the year.

The aforementioned data aim to investigate the rhinitis and dysphagia symptoms of the patients in the last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All the subjects with EOE diagnosis

Exclusion Criteria:

* All the patients without EOE diagnosis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the subjects (both sex) between 18 and 75 years old with EOE diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the recrudescence of dysphagia symptoms and Seasons | 12 months
  Evaluate the possible correlation between the recrudescence of dysphagia symptoms and a specific month of the year and/or specific season.

SECONDARY OUTCOMES:
Correlation between the anamnestic onset of the disease and the individual patient's sensitization to aeroallergens. | 12 months
  Evaluate whether there is a statistically significant correlation between the anamnestic onset of the disease and the individual patient's sensitization to aeroallergens.
Prevalence of respiratory allergy (rhinitis and allergic asthma) in patients with EoE. | 12 months
  Evaluate the prevalence of respiratory allergy (rhinitis and allergic asthma) in patients with EoE.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy